CLINICAL TRIAL: NCT03863925
Title: Comparison of Propofol Target-Controlled Infusion Anesthesia and Bolus Injection in Electroconvulsive Therapy: A Randomized Controlled Trial
Brief Title: Comparison of Propofol Target-Controlled Infusion Anesthesia and Bolus Injection in Electroconvulsive Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201700862A3
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2017-08

CONDITIONS: Depression; Schizophrenia; Bipolar Disorder; Cognitive Dysfunction
Keywords: Electroconvulsive therapy; Propofol; Target controlled infusion
MeSH Terms: conditions — Depression; Schizophrenia; Bipolar Disorder; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol Target Controlled Infusion Group (Group T) (Experimental): Patients in group T underwent anesthesia with Propofol (dosage form: 10mg/mL) target controlled infusion by Schnider model, starting at concentration of effect site (Ce) of 1.5 mcg/mL and titrating to achieve Observer's Assessment of Alertness/Sedation (OAA/S) Scale level 3 (responds only after name called loudly or repeatedly). Patients were paralyzed with suxamethonium (dosage form: 20mg/mL; dosage: 1mg/kg) once adequate sedation level achieved. TCI was stopped once the psychiatrist applied electroconvulsive stimulation to patients' bilateral frontal regions. Assisted ventilation with bag-valve-mask device by experienced anesthesiologists was began since patients were sedated until adequate spontaneous respiration was regained after each single electroconvulsive therapy (ECT) session. Every patient receive total six to twelve ECT sessions, and each ECT session was conducted one day apart.
  Interventions: Device: Target controlled infusion, Schnider model
- Propofol Bolus Group (Group B) (Active Comparator): Patients in group B underwent anesthesia with bolus of propofol for sedation, and the dosage raged between 0.75 to 1.5 mg/kg to achieve at least OAA/S scale level 3. Dosage of suxamethonium, application of electroconvulsive stimulation, ventilation maneuver, frequency of ECT session, and number of total ECT sessions were same as patients in group T.
  Interventions: Behavioral: Bolus injection of Propofol

INTERVENTIONS:
Device: Target controlled infusion, Schnider model — Target controlled infusion (TCI) is an intravenous drug delivery system estimating pharmacokinetics after input of patient's data, e.g. age, sex, body height, body weight. Schnider model is one of TCI model to deliver Propofol. After target concentration at effect site (e.g. the brain) is keyed in, the computerized infusion pump will calculate dosage of bolus and infusion rate for each individual, and calculated concentration of propofol at plasma and brain will be displayed. The clinicians should evaluate the patient's sedation level in response to calculated propofol concentration and titrate target concentration to achieve desired sedation level.
  Arms: Propofol Target Controlled Infusion Group (Group T)
Behavioral: Bolus injection of Propofol — Bolus intravenous injection is a traditional way to deliver anesthetic, and the dosage and amount of medication is based on clinical experience and patients' response.
  Arms: Propofol Bolus Group (Group B)

SUMMARY:
Electroconvulsive therapy (ECT) serves as an effective adjuvant or alternative modality for major depressive disorder, schizophrenia, or bipolar affective disorder refractory to or contraindicated to psychopharmacological treatment. Anesthetics have been introduced into ECT sessions to alleviate ECT-inducing discomfort sensation, tachycardia, arrhythmia, hypertension, and anxiety. Propofol is highly lipid soluble and able to rapidly cross the blood-brain barrier (BBB), which leads to rapid onset of sedation and hypnosis. Meanwhile, propofol has hemodynamic depressant effect and attenuates hypertensive surge during ECT. Characteristics mentioned above make propofol one of widely used anesthetics for anesthetized ECT.

Propofol can be administered with bolus injection or target-controlled infusion (TCI). Compared with bolus injection, TCI provides relatively constant concentration at site of interest based on computer simulation with input of pharmacokinetic parameters, such as age, body weight, body height, etc. However, propofol is also well known for anticonvulsant property, which may inevitably interfere with seizure propagation by electroconvulsive stimulus and diminish consequent efficacy. Thus, dosage of electrical stimulus may be increased to achieve ideal seizure quality in this setting, which also leads to higher risk of subsequent cognitive impairment.

In our clinical practice, TCI system reduces total amount of propofol in comparison with bolus injection method. Therefore, we hypothesize that application of TCI system in anesthetized ECT relates to lower dosage of electrical stimulus and decreased incidence or severity of post-treatment cognitive impairment.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) serves as an effective adjuvant or alternative modality for major depressive disorder, schizophrenia, or bipolar affective disorder refractory to or contraindicated to psychopharmacological treatment. Anesthetics have been introduced into ECT sessions to alleviate ECT-inducing discomfort sensation, tachycardia, arrhythmia, hypertension, and anxiety. Propofol is highly lipid soluble and able to rapidly cross the blood-brain barrier (BBB), which leads to rapid onset of sedation and hypnosis. Meanwhile, propofol has hemodynamic depressant effect and attenuates hypertensive surge during ECT. Characteristics mentioned above make propofol one of widely used anesthetics for anesthetized ECT.

Propofol can be administered with bolus injection or target-controlled infusion (TCI). Compared with bolus injection, TCI provides relatively constant concentration at site of interest based on computer simulation with input of pharmacokinetic parameters, such as age, body weight, body height, etc. However, propofol is also well known for anticonvulsant property, which may inevitably interfere with seizure propagation by electroconvulsive stimulus and diminish consequent efficacy. Thus, dosage of electrical stimulus may be increased to achieve ideal seizure quality in this setting, which also leads to higher risk of subsequent cognitive impairment.

In our clinical practice, TCI system reduces total amount of propofol in comparison with bolus injection method. Therefore, we hypothesize that application of TCI system in anesthetized ECT relates to lower dosage of electrical stimulus and decreased incidence or severity of post-treatment cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 years old and 65 years old
* Diagnosis of major depressive disorder, bipolar disorder, and schizophrenia, compatible with SCID for DSM-5, with clinical necessity of ECT under a psychiatrist's evaluation and decision
* Patients with adequate visual acuity and auditory acuity without or with correction
* Patients or patients' legal representative signing up the informed consent

Exclusion Criteria:

* Patients already diagnosed with neurocognitive disorder
* Patients with contraindications to ECT, including myocardial infarction, cerebrovascular disease, elevated intracranial pressure, intracranial angiomas, untreated bony fractures, cervical spine injury, pheochromocytoma, heart failure, sever valvular disease, deep vein thrombosis, etc.
* Patients with untreated substance abuse, including alcohol and illegal drugs
* Patients with unspecified psychiatric disorders
* Patients unable to cooperate

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline Clinical Global Impression-Severity (CGI-S) | through study completion, an average of one month
  Evaluation with Clinical Global Impression-Severity (CGI-S)
Change from baseline Clinical Global Impression-Improvement (CGI-I) | through study completion, an average of one month
  Evaluation with Clinical Global Impression-Improvement (CGI-I)

SECONDARY OUTCOMES:
Cognitive dysfunction | through study completion, an average of one month
  Evaluation with Montreal Cognitive Assessment (MoCA)

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ling Hsieh, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Semkovska M, McLoughlin DM. Objective cognitive performance associated with electroconvulsive therapy for depression: a systematic review and meta-analysis. Biol Psychiatry. 2010 Sep 15;68(6):568-77. doi: 10.1016/j.biopsych.2010.06.009. Epub 2010 Jul 31. PMID 20673880
- [Background] Sackeim HA, Prudic J, Fuller R, Keilp J, Lavori PW, Olfson M. The cognitive effects of electroconvulsive therapy in community settings. Neuropsychopharmacology. 2007 Jan;32(1):244-54. doi: 10.1038/sj.npp.1301180. Epub 2006 Aug 23. PMID 16936712
- [Background] McClintock SM, Choi J, Deng ZD, Appelbaum LG, Krystal AD, Lisanby SH. Multifactorial determinants of the neurocognitive effects of electroconvulsive therapy. J ECT. 2014 Jun;30(2):165-76. doi: 10.1097/YCT.0000000000000137. PMID 24820942
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Sakamoto A, Hoshino T, Suzuki N, Suzuki H, Kimura M, Ogawa R. Effects of propofol anesthesia on cognitive recovery of patients undergoing electroconvulsive therapy. Psychiatry Clin Neurosci. 1999 Dec;53(6):655-60. doi: 10.1046/j.1440-1819.1999.00621.x. PMID 10687746
- [Background] Imashuku Y, Kanemoto K, Senda M, Matsubara M. Relationship between blood levels of propofol and recovery of memory in electroconvulsive therapy. Psychiatry Clin Neurosci. 2014 Apr;68(4):270-4. doi: 10.1111/pcn.12122. Epub 2013 Dec 8. PMID 24313665
- [Background] Galvez V, Hadzi-Pavlovic D, Wark H, Harper S, Leyden J, Loo CK. The Anaesthetic-ECT Time Interval in Electroconvulsive Therapy Practice--Is It Time to Time? Brain Stimul. 2016 Jan-Feb;9(1):72-7. doi: 10.1016/j.brs.2015.09.005. Epub 2015 Sep 12. PMID 26452698
- [Background] Struys MM, De Smet T, Glen JI, Vereecke HE, Absalom AR, Schnider TW. The History of Target-Controlled Infusion. Anesth Analg. 2016 Jan;122(1):56-69. doi: 10.1213/ANE.0000000000001008. PMID 26516804
- [Derived] Hsieh ML, Lu YT, Lin CC, Lee CP. Comparison of the target-controlled infusion and the manual infusion of propofol anesthesia during electroconvulsive therapy: an open-label randomized controlled trial. BMC Psychiatry. 2021 Feb 4;21(1):71. doi: 10.1186/s12888-021-03069-6. PMID 33541306